CLINICAL TRIAL: NCT04680832
Title: Exhaled Breath Analysis Using eNose Technology as a Biomarker for Diagnosis and Disease Progression in Fibrotic Interstitial Lung Disease
Brief Title: Exhaled Breath Analysis Using eNose Technology as a Biomarker for Diagnosis and Disease Progression in Fibrotic ILD
Acronym: ILDnose
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Principal Investigator, MD PhD, Erasmus Medical Center
Other Study IDs: MEC-2020-0655
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ILD patients: Patients diagnosed with one of the most prevalent fibrotic ILDs: IPF, CHP, CTD-ILD, iNSIP, IPAF, and unclassifiable ILD (defined as unclassifiable disease at the time of the first MDT).
  Interventions: Diagnostic Test: Electronic nose

INTERVENTIONS:
Diagnostic Test: Electronic nose — First, patients will be asked to rinse their mouth thoroughly with water three times. Subsequently, exhaled breath analysis will be performed in duplicate with a 1-minute interval. An eNose measurement consists of five tidal breaths, followed by an inspiratory capacity maneuver to total lung capacity, a five second breath hold, and subsequently a slow expiration (flow <0.4L/s) to residual volume. The measurements are non-invasive and will cost approximately 5-10 minutes in total, including explanation and informed consent procedure. There are no risks associated with this study and the burden for patients is minimal.
  Other Names: SpiroNose; eNose

SUMMARY:
The ILDnose study a multinational, multicenter, prospective, longitudinal study in outpatients with pulmonary fibrosis. The aim is to assess the accuracy of eNose technology as diagnostic tool for diagnosis and differentiation between the most prevalent fibrotic interstitial lung diseases. The value of eNose as biomarker for disease progression and response to treatment is also assessed. Besides, validity of several questionnaires for pulmonary fibrosis is investigated.

DETAILED DESCRIPTION:
Patients will be included in the study after signing written informed consent. eNose measurements will take place before or after a routine outpatient clinic visit at the same location as the regular visit, ensuring minimal inconvenience for patients. First, patients will be asked to rinse their mouth thoroughly with water three times. Subsequently, exhaled breath analysis will be performed in duplicate with a 1-minute interval. An eNose measurement consists of five tidal breaths, followed by an inspiratory capacity maneuver to total lung capacity, a five second breath hold, and subsequently a slow expiration (flow <0.4L/s) to residual volume. The measurements are non-invasive and will cost approximately 5-10 minutes in total, including explanation and informed consent procedure. There are no risks associated with this study and the burden for patients is minimal.

After the measurement, patients will complete a short survey about questions relevant for the data analysis (food intake in the last two hours, smoking history, medication use, comorbidities, and symptoms of respiratory infection). In addition, patients will complete the L-PF questionnaire and the Global Rating of Change scale (GRoC). The L-PF questionnaire consists of 21 questions on a 5-point Likert scale about the impact of pulmonary fibrosis on quality of life, and takes about 3 minutes to complete. The GRoC consists of one question on a scale from -7 to 7: were there any changes in your quality of life since your last visit? Symptoms (cough and dyspnea) will be scored on a 10 cm VAS scale from -5 to 5.

Next to eNose measurements, demographic data and physiological parameters of patients will be collected from the medical records at baseline, month 6, and month 12. Parameters such as age, gender, diagnosis, time since diagnosis, comorbidities, medication, pulmonary function (forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO)), laboratory parameters (i.e. auto-immune antibodies), HRCT pattern, BAL results and if applicable also genetic mutations, will be recorded and stored in an electronic case report form. These parameters will be collected as part of routine daily care, patients will not undergo any additional tests for study purposes. HRCT scans will be re-analysed centrally by an experienced ILD thoracic radiologist. Mortality and lung function parameters will also be collected at 24 months, if this information is available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of fibrotic ILD, as discussed in a multidisciplinary team meeting (50% incident patients and 50% prevalent patients). Patients are classified as 'incident' if they received a diagnosed in a multidisciplinary team meeting within the past six months. Patients will be required to have fibrosis on a HRCT scan <1 year before enrollment in the study defined as reticular abnormality with traction bronchiectasis, with or without honeycombing, as determined by a radiologist. No minimum extent of fibrosis will be required.

Exclusion Criteria:

* Alcohol consumption ≤ 12 hours before the measurement
* Physically not able to perform eNose measurement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ILD
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for IPF - CHP | Baseline
  Accuracy for differentiating IPF from CHP
AUC for IPF - CHP | Baseline
  AUC for differentiating IPF from CHP
AUC for IPF - iNSIP | Baseline
  AUC for differentiating IPF from iNSIP
Diagnostic accuracy for IPF - iNSIP | Baseline
  Accuracy for differentiating IPF from iNSIP
AUC for IPF - IPAF | Baseline
  AUC for differentiating IPF from IPAF
Diagnostic accuracy for IPF - IPAF | Baseline
  Accuracy for differentiating IPF from IPAF
Diagnostic accuracy for IPF - CTD-ILD | Baseline
  Accuracy for differentiating IPF from CTD-ILD
AUC for IPF - CTD-ILD | Baseline
  AUC for differentiating IPF from CTD-ILD
Diagnostic accuracy for IPF - unclassifiable ILD | Baseline
  Accuracy for differentiating IPF from unclassifiable ILD
AUC for IPF - unclassifiable ILD | Baseline
  AUC for differentiating IPF from unclassifiable ILD
Diagnostic accuracy for CHP - iNSIP | Baseline
  Accuracy for differentiating CHP from iNSIP
AUC for CHP - iNSIP | Baseline
  AUC for differentiating CHP from iNSIP
Diagnostic accuracy for CHP - IPAF | Baseline
  Accuracy for differentiating CHP from IPAF
AUC for CHP - IPAF | Baseline
  AUC for differentiating CHP from IPAF
Diagnostic accuracy for CHP - CTD-ILD | Baseline
  Accuracy for differentiating CHP from CTD-ILD
AUC for CHP - CTD-ILD | Baseline
  AUC for differentiating CHP from CTD-ILD
Diagnostic accuracy for CHP - unclassifiable ILD | Baseline
  Accuracy for differentiating CHP from unclassifiable ILD
AUC for CHP - unclassifiable ILD | Baseline
  AUC for differentiating CHP from unclassifiable ILD
Diagnostic accuracy for iNSIP - IPAF | Baseline
  Accuracy for differentiating iNSIP from IPAF
AUC for iNSIP - IPAF | Baseline
  AUC for differentiating iNSIP from IPAF
Diagnostic accuracy for iNSIP - CTD-ILD | Baseline
  Accuracy for differentiating iNSIP from CTD-ILD
AUC for iNSIP - CTD-ILD | Baseline
  AUC for differentiating iNSIP from CTD-ILD
Diagnostic accuracy for iNSIP - unclassifiable ILD | Baseline
  Accuracy for differentiating iNSIP from unclassifiable ILD
AUC for iNSIP - unclassifiable ILD | Baseline
  AUC for differentiating iNSIP from unclassifiable ILD
Diagnostic accuracy for IPAF - CTD-ILD | Baseline
  Accuracy for differentiating IPAF from CTD-ILD
AUC for IPAF - CTD-ILD | Baseline
  AUC for differentiating IPAF from CTD-ILD
Diagnostic accuracy for IPAF - unclassifiable ILD | Baseline
  Accuracy for differentiating IPAF from unclassifiable ILD
AUC for IPAF - unclassifiable ILD | Baseline
  AUC for differentiating IPAF from unclassifiable ILD
Diagnostic accuracy for CTD-ILD - unclassifiable ILD | Baseline
  Accuracy for differentiating CTD-ILD from unclassifiable ILD
AUC for CTD-ILD - unclassifiable ILD | Baseline
  AUC for differentiating CTD-ILD from unclassifiable ILD
Disease progression | 12 months after inclusion
  FVC decline in combination with worsening of respiratory symptoms (cough and/or dyspnea) and/or progressive fibrosis on CT scan
Disease progression | 24 months after inclusion
  FVC decline in combination with worsening of respiratory symptoms (cough and/or dyspnea) and/or progressive fibrosis on CT scan
Diagnostic accuracy of disease progression | 6 months after inclusion
  Relating disease progression (based on FVC decline, CT scan and/or symptoms) to change in eNose values
Diagnostic accuracy of disease progression | 12 months after inclusion
  Relating disease progression (based on FVC decline, CT scan and/or symptoms) to change in eNose values
Diagnostic accuracy of disease progression | 24 months after inclusion
  Relating disease progression (based on FVC decline, CT scan and/or symptoms) to change in eNose values
Worsening of respiratory symptoms (cough and/or dyspnea) | 12 months after inclusion
  Worsening of respiratory symptoms (cough and/or dyspnea) measured on a visual analogue scale (0-10, 0 no symptoms, 10 most severe symptoms)
Mortality | 12 months after inclusion
  Deceased subjects
Mortality | 24 months after inclusion
  Deceased subjects
Therapeutic effect | 6 months after start therapy
  Relating start of anti-fibrotic medication to change in eNose values
Therapeutic effect | 12 months after start therapy
  Relating start of anti-fibrotic medication to change in eNose values

SECONDARY OUTCOMES:
L-PF evaluation | 6 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to eNose values
L-PF evaluation | 6 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to lung function values
L-PF evaluation | 12 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to eNose values
L-PF evaluation | 12 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to lung function values
L-PF evaluation | 24 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to eNose values
L-PF evaluation | 24 months after inclusion
  Relating Longitudinal changes in score of L-PF questionnaire to lung function values
GRoC evaluation | 6 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to eNose values
GRoC evaluation | 6 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to lung function values
GRoC evaluation | 12 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to eNose values
GRoC evaluation | 12 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to lung function values
GRoC evaluation | 24 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to eNose values
GRoC evaluation | 24 months after inclusion
  Relating Longitudinal changes in score of Global Rating of Change Scale to lung function values

CONTACTS AND LOCATIONS:
Overall Officials: Marlies S Wijsenbeek, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- University Lyon 1, Louis Pradel hospital, Lyon. FranceService de pneumologie, hôpital Louis Pradel, Lyon, France
- Thoraxklinik Heidelberg, Heidelberg, Germany
- Erasmus MC, Rotterdam, Netherlands
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No